CLINICAL TRIAL: NCT03910244
Title: Pomalidomide for the Treatment of Bleeding in Hereditary Hemorrhagic Telangiectasia
Brief Title: Pomalidomide for the Treatment of Bleeding in HHT
Acronym: PATH-HHT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: RTI International (Other)
Responsible Party: Principal Investigator, Keith McCrae, Director, Benign Hematology, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 133646
Record Dates: First submitted 2019-04-08; First posted 2019-04-10 (Actual); Results first posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-09

CONDITIONS: Telangiectasia, Hereditary Hemorrhagic
Keywords: Epistaxis; pomalidomide; blood transfusion
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic; Epistaxis | interventions — pomalidomide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pomalidomide (Experimental): Oral Pomalidomide will be provided as a capsule at 4 mg/day dose. There will be 6 treatment cycles of 28 days (4 weeks) each. Total treatment phase duration will be 24 weeks.
  Interventions: Drug: Pomalidomide Oral Product
- Placebo (Placebo Comparator): A placebo matching the study drug will be provided as a capsule. There will be 6 treatment cycles of 28 days (4 weeks) each. Total treatment phase duration will be 24 weeks.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Pomalidomide Oral Product — Pomalidomide, a third generation derivative of thalidomide, given orally at a starting dose of 4 mg/day for days 1-28 of six 28-day cycles. The dose may be reduced to 3 or 2 mg/day based on specific adverse event (AE) criteria.
  Other Names: POMALYST
  Arms: Pomalidomide
Drug: Placebo oral capsule — Matching placebo will be given.
  Arms: Placebo

SUMMARY:
This is a Phase II placebo-controlled double-blind study of pomalidomide in patients with hereditary hemorrhagic telangiectasia (HHT) with moderate to severe epistaxis who have anemia and/or require parenteral iron infusions or blood transfusions. A total of 159 patients will be randomized 2:1 to treatment with oral pomalidomide or matching placebo for 24 weeks. Mean change from baseline to 24 weeks in the Epistaxis Severity Score (ESS) will be compared between treatment groups to determine pomalidomide efficacy.

DETAILED DESCRIPTION:
HHT is associated with substantial morbidity, leading to a reduced quality of life, decreased rate of employment and a high incidence of depression. There currently exists no medical therapy recognized as consistently efficacious in HHT. Reports of the efficacy of thalidomide in HHT, as well as interim results of a pilot trial of pomalidomide in HHT provide evidence of efficacy with minimal toxicity. The favorable efficacy:toxicity ratio of pomalidomide suggest that it may benefit patients with HHT.

This study is designed as a Phase II placebo-controlled double-blind study of pomalidomide in HHT patients with moderate to severe epistaxis who have anemia and/or require parenteral iron infusions or blood transfusions. A total of 159 patients will be randomized 2:1 to treatment with oral pomalidomide or matching placebo for 24 weeks.

Primary Objective: To determine efficacy of pomalidomide compared to placebo for the reduction in severity of epistaxis after 24 weeks of treatment.

Secondary Objectives: To determine the safety and tolerability of pomalidomide for the treatment of HHT; to determine if pomalidomide treatment improves quality of life in HHT; to determine whether a continued response to pomalidomide is evident 4 weeks after treatment discontinuation; to develop a biorepository for future studies to define biomarkers predictive of pomalidomide response and allow investigations into the biology of HHT and mechanisms of pomalidomide.

ELIGIBILITY:
Inclusion Criteria:

1. A clinical diagnosis of HHT as defined by the Curacao criteria
2. Age ≥ 18 years
3. Platelet count ≥ 100,000/µl
4. White Blood Count (WBC) ≥ 2,500/µl
5. International Normalized Ratio (INR) ≤ 1.4 and normal ± 2 sec activated partial thromboplastin time (aPTT or partial thromboplastin time (PTT) per local laboratory designation) by local laboratory criteria (except for patients on a stable dose of warfarin or direct oral anticoagulants)
6. Epistaxis severity score ≥ 3 measured over the preceding three months, measured at the screening visit
7. A requirement for anemia, as determined by local laboratory hemoglobin assessment and normal ranges, and/or parenteral infusion of at least 250 mg of iron or transfusion of 1 unit of blood over the 24 weeks preceding the screening visit
8. All study participants must agree to be registered into the FDA mandated POMALYST Risk Evaluation and Mitigation Strategy (REMS) program, and be willing and able to comply with the requirements of the POMALYST REMS program
9. Females of childbearing potential (FCBP) must adhere to the scheduled pregnancy testing as required in the POMALYST REMS program. FCBP must have a negative pregnancy test with a sensitivity of at least 50 milli-international units per milliliter (mIU/mL) within 10 - 14 days prior to and again within 24 hours prior to prescribing pomalidomide and must either commit to continued abstinence from heterosexual intercourse or use two (2) acceptable methods of birth control, one highly effective method and one additional effective method at the same time, at least 28 days before she starts taking pomalidomide, during therapy and for at least 4 weeks following discontinuation of therapy. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a vasectomy.
10. Ability to understand and sign informed consent

Exclusion Criteria:

1. Women currently breast feeding
2. Renal insufficiency, serum creatinine > 2.0 mg/dl
3. Hepatic insufficiency, bilirubin > 2.0 (or >4.0 in the setting of a prior clinical or genetic diagnosis of Gilbert's syndrome) or transaminases > 3.0x normal
4. Prior treatment with thalidomide or other Immunomodulatory imide drugs within previous 6 months
5. Prior treatment with bevacizumab (systemic or nasal) within previous 6 weeks*
6. Prior treatment with pazopanib within previous 6 weeks*
7. The use of octreotide or oral estrogens within the previous month*
8. History of prior unprovoked thromboembolism confirmed by venous ultrasound or other imaging modalities
9. Peripheral neuropathy, confirmed by neurologic consultation
10. Known underlying hypoproliferative anemia (i.e. myelodysplasia, aplastic anemia)
11. Currently enrolled in other interventional trials
12. Known hypersensitivity to thalidomide or lenalidomide.
13. The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
14. Known SMAD Family Member 4 (SMAD-4) mutation, unless there has been a colonoscopy with normal (negative) results, or in which the patient has had no more than 5 small (in the opinion of the gastroenterologist) colonic polyps completely removed within the preceding 18 months
15. Anything that in the investigator's opinion is likely to interfere with completion of the study

    * * Use of these treatments is not permitted during study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2019-10-17 (Actual); Primary Completion 2023-09-08 (Actual); Study Completion 2023-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith McCrae, MD, Principal Investigator — The Cleveland Clinic
Locations (14):
- United States (14):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - UCSD Hemophilia and Thrombosis Treatment Center, San Diego, California
  - UCSF Outpatient Hematology Clinic, San Francisco, California
  - University of Florida, Gainesville, Florida
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Massachussets General Hospital, Boston, Massachusetts
  - University of Minnesota Health Clinical Research Unit, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of North Carolina, Chapel Hill, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania Perelman School of Medicine, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Texas Children's Hospital, Houston, Texas
  - University of Utah Healthcare, Salt Lake City, Utah
  - Medical College of Wiconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
The Data Coordinating Center (DCC) will prepare de-identified data files for sharing. A final data sharing plan will be developed with NHLBI and the study Steering Committee (SC). The data can be provided in Statistical Analysis System (SAS) data sets and export files and documentation will be in portable document format (PDF).
  The first level of data sharing will be with trial investigators. In addition, the DCC will be responsible for sharing study data with outside researchers, if approved by NHLBI and the SC.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be made available to investigators 6 months after closed data sets for the trial have been prepared for final analysis or 1 month after results of the protocol are published in a peer-reviewed journal.
Access Criteria: A data request form will be developed to collect information deemed necessary by the SC and NIH, including applicant name, organization, and purpose of research. Investigators will submit the request form, Data Distribution Agreement, and Institutional Review Board (IRB) approval to designated DCC staff. The SC or its designated Committee will review each application, and if the requestor meets established criteria for access to the data and provides the required documents, the requested data sets and associated documentation will be disseminated by a mode agreed upon by the SC in accordance with NHLBI policy.

REFERENCES:
- [Background] McDonald J, Wooderchak-Donahue W, VanSant Webb C, Whitehead K, Stevenson DA, Bayrak-Toydemir P. Hereditary hemorrhagic telangiectasia: genetics and molecular diagnostics in a new era. Front Genet. 2015 Jan 26;6:1. doi: 10.3389/fgene.2015.00001. eCollection 2015. PMID 25674101
- [Background] Hoag JB, Terry P, Mitchell S, Reh D, Merlo CA. An epistaxis severity score for hereditary hemorrhagic telangiectasia. Laryngoscope. 2010 Apr;120(4):838-43. doi: 10.1002/lary.20818. PMID 20087969
- [Background] Chaturvedi S, Clancy M, Schaefer N, Oluwole O, McCrae KR. Depression and post-traumatic stress disorder in individuals with hereditary hemorrhagic telangiectasia: A cross-sectional survey. Thromb Res. 2017 May;153:14-18. doi: 10.1016/j.thromres.2017.03.003. Epub 2017 Mar 9. PMID 28314138
- [Derived] Al-Samkari H, Kasthuri RS, Iyer VN, Pishko AM, Decker JE, Weiss CR, Whitehead KJ, Conrad MB, Zumberg MS, Zhou JY, Parambil J, Marsh D, Clancy M, Bradley L, Wisniewski L, Carper BA, Thomas SM, McCrae KR. Pomalidomide for Epistaxis in Hereditary Hemorrhagic Telangiectasia. N Engl J Med. 2024 Sep 19;391(11):1015-1027. doi: 10.1056/NEJMoa2312749. PMID 39292928

RESULTS

PARTICIPANT FLOW:
Groups:
- Pomalidomide: Daily dose of 4, 3, or 2 mg of Pomalidomide for 24 weeks
- Placebo: Daily dose of placebo for 24 weeks
Period: Overall Study
Arm/Group | Pomalidomide | Placebo
Started | 95 | 49
Completed | 63 | 41
Not Completed | 32 | 8
Not completed — Adverse Event | 14 | 0
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 0 | 2
Not completed — Joint withdrawal decision | 1 | 0
Not completed — Study Terminated by Sponsor | 7 | 4
Not completed — Physician Decision | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 7 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Pomalidomide | Total
Number analyzed (Participants) | 49 | 95 | 144
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.7 (11) | 58.8 (13) | 58.8 (12)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 24 | 45 | 69
  Male | 25 | 50 | 75
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 0 | 1
  Black/African American | 5 | 6 | 11
  Other | 0 | 3 | 3
  Unknown | 2 | 1 | 3
  White | 41 | 85 | 126
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic/Latino | 3 | 2 | 5
  Not Hispanic/Latino | 44 | 90 | 134
  Unknown/Not Reported | 2 | 3 | 5
Marital status [Count of Participants; unit: Participants]
  Divorced | 3 | 10 | 13
  Domestic Partner | 0 | 2 | 2
  Married | 33 | 64 | 97
  Never Been Married | 9 | 15 | 24
  Separated | 2 | 1 | 3
  Unknown | 0 | 1 | 1
  Widowed | 2 | 2 | 4
Pre-menopausal [Count of Participants; unit: Participants]
  No | 17 | 33 | 50
  Not Applicable | 25 | 50 | 75
  Yes | 7 | 12 | 19
Education [Count of Participants; unit: Participants]
  Associate degree | 5 | 8 | 13
  Bachelor�s degree | 12 | 15 | 27
  Doctoral degree | 1 | 5 | 6
  Don�t Know | 18 | 36 | 54
  High School Grad | 4 | 9 | 13
  Master�s degree | 4 | 9 | 13
  Refused | 1 | 3 | 4
  Years of college no degree (specify) | 4 | 9 | 13
  grade (specify) | 0 | 1 | 1
Employment status [Count of Participants; unit: Participants]
  Disabled permanently or temporary | 3 | 2 | 5
  Looking for work unemployed | 0 | 1 | 1
  Other (specify) | 9 | 16 | 25
  Retired | 12 | 28 | 40
  Working Now | 25 | 48 | 73
Emergency room for epistaxis in the previous 3 months [Count of Participants; unit: Participants]
  No | 40 | 79 | 119
  Yes | 9 | 16 | 25
History of or current GI bleeding [Count of Participants; unit: Participants]
  No | 30 | 61 | 91
  Yes | 19 | 34 | 53
HHT involvement of the brain [Count of Participants; unit: Participants]
  No | 39 | 77 | 116
  Unknown | 4 | 9 | 13
  Yes | 6 | 9 | 15
HHT involvement of the liver [Count of Participants; unit: Participants]
  No | 28 | 47 | 75
  Unknown | 11 | 23 | 34
  Yes | 10 | 25 | 35
HHT involvement of the lungs [Count of Participants; unit: Participants]
  No | 25 | 45 | 70
  Unknown | 8 | 8 | 16
  Yes | 16 | 42 | 58
HHT Diagnosis Genetically Confirmed [Count of Participants; unit: Participants]
  No | 3 | 7 | 10
  Yes | 46 | 88 | 134
Endoglin Gene (ENG) Mutation [Count of Participants; unit: Participants]
  Known Pathogenic Mutation | 13 | 35 | 48
  No Mutation | 8 | 16 | 24
  Not done | 4 | 8 | 12
  Unknown | 23 | 33 | 56
  Variant of Unknown Significanc | 1 | 1 | 2
  Variant, Likely Pathogenic | 0 | 2 | 2
Activin A Receptor Like Type 1 Gene (ACVRL1) Mutation [Count of Participants; unit: Participants]
  Known Pathogenic Mutation | 25 | 34 | 59
  No Mutation | 5 | 8 | 13
  Not done | 3 | 10 | 13
  Unknown | 8 | 30 | 38
  Variant of Unknown Significanc | 2 | 9 | 11
  Variant, Likely Pathogenic | 6 | 4 | 10
SMAD4 Mutation [Count of Participants; unit: Participants]
  Known Pathogenic Mutation | 0 | 1 | 1
  No Mutation | 10 | 20 | 30
  Not done | 6 | 13 | 19
  Unknown | 33 | 61 | 94
EPHB4 Mutation [Count of Participants; unit: Participants]
  No Mutation | 10 | 12 | 22
  Not done | 6 | 21 | 27
  Unknown | 33 | 62 | 95
Growth Differentiation Factor 2 (GDF2) Mutation [Count of Participants; unit: Participants]
  No Mutation | 10 | 16 | 26
  Not done | 6 | 17 | 23
  Unknown | 33 | 62 | 95
RAS p21 Protein Activator (RASA1) Mutation [Count of Participants; unit: Participants]
  No Mutation | 10 | 16 | 26
  Not done | 6 | 17 | 23
  Unknown | 33 | 61 | 94
  Variant of Unknown Significanc | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Epistaxis Severity Score
Description: The primary outcome measure is the change from baseline in Epistaxis Severity Score (ESS) after 6 months of treatment administration to compare the outcomes of Pomalidomide versus Placebo. The ESS ranges from 0-10 with higher scores indicating worse condition in the prior 4 weeks. The minimal important difference is 0.71
Time Frame: 4, 8, 12, 16, 20, and 24 Weeks and 4 weeks post treatment
Population: An intent-to-treat (ITT) analysis which included all randomized participants who provided outcome data.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 49 | 92
units on a scale
  4 Weeks | -1 [-1.40 to -0.60] | -1.1 [-1.50 to -0.70]
  8 Weeks: number analyzed (Participants) | 49 | 87
  8 Weeks | -1.3 [-1.80 to -0.70] | -1.2 [-1.60 to -0.80]
  12 Weeks: number analyzed (Participants) | 46 | 77
  12 Weeks | -1.3 [-1.90 to -0.80] | -1.6 [-2.00 to -1.20]
  16 Weeks: number analyzed (Participants) | 44 | 73
  16 Weeks | -1.2 [-1.90 to -0.60] | -2 [-2.40 to -1.60]
  20 Weeks: number analyzed (Participants) | 43 | 66
  20 Weeks | -1.3 [-1.90 to -0.60] | -2 [-2.40 to -1.50]
  24 Weeks: number analyzed (Participants) | 43 | 63
  24 Weeks | -1.2 [-1.90 to -0.50] | -2.1 [-2.60 to -1.50]
  4 Weeks Post-treatmenr: number analyzed (Participants) | 41 | 63
  4 Weeks Post-treatmenr | -0.7 [-1.30 to 0.00] | -1.6 [-2.10 to -1.20]

2. Secondary Outcome: Average Total Daily Duration of Nosebleeds - Change From Baseline
Description: The daily epistaxis duration is calculated as the total duration of all reported nose bleeding events in a day, averaged across all days reported in a 4-week smartphone diary. The outcome is the change between the baseline diary on the specified timepoint
Time Frame: After 12 and 24 weeks of treatment, and 4 weeks post-treatment
Population: An intent-to-treat (ITT) analysis which included all randomized participants who provided outcome data.
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 43 | 73
minutes
  12 Weeks: number analyzed (Participants) | 35 | 64
  12 Weeks | -4 [-8.40 to 0.50] | -6.7 [-10.40 to -3.00]
  24 Weeks: number analyzed (Participants) | 32 | 53
  24 Weeks | -4.4 [-10.50 to 1.70] | -5.3 [-11.00 to 0.50]
  4 Weeks Post-treatment: number analyzed (Participants) | 31 | 49
  4 Weeks Post-treatment | -1.7 [-7.50 to 4.20] | -4.6 [-7.90 to -1.30]

3. Secondary Outcome: Weighted Average Total Daily Duration of Nosebleeds - Change From Baseline
Description: The daily epistaxis duration is calculated as the total duration of all reported nose bleeding events in a day, averaged across all days reported in a 4-week smartphone diary, weighted by the intensity, with 90%% winsorization. The outcome is the change between the baseline diary on the specified timepoint
Time Frame: After 12 and 24 weeks of treatment, and 4 weeks post-treatment
Population: An intent-to-treat (ITT) analysis which included all randomized participants who provided outcome data.
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 43 | 73
minutes
  12 Weeks: number analyzed (Participants) | 35 | 64
  12 Weeks | -4.3 [-10.40 to 1.70] | -12.1 [-16.60 to -7.60]
  24 Weeks: number analyzed (Participants) | 32 | 53
  24 Weeks | -4 [-13.50 to 5.60] | -11.5 [-16.60 to -6.30]
  4 Weeks Post-treatment: number analyzed (Participants) | 31 | 49
  4 Weeks Post-treatment | -2.6 [-10.60 to 5.40] | -9.3 [-14.10 to -4.60]

4. Other Pre Specified Outcome: Average Total Daily Duration of Low Intensity Nosebleeds - Change From Baseline
Description: The daily of low intensity epistaxis duration is calculated as the total duration of "spotting" or "dripping" nose bleeding events in a day, averaged across all days reported in a 4-week smartphone diary. The outcome is the change between the baseline diary on the specified timepoint
Time Frame: After 12 and 24 weeks of treatment, and 4 weeks post-treatment
Population: An intent-to-treat (ITT) analysis which included all randomized participants who provided outcome data.
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 43 | 73
minutes
  12 Weeks: number analyzed (Participants) | 35 | 64
  12 Weeks | -2 [-5.20 to 1.30] | -1.6 [-2.90 to -0.20]
  24 Weeks: number analyzed (Participants) | 32 | 53
  24 Weeks | -2.8 [-6.10 to 0.50] | -1.6 [-2.70 to -0.40]
  4 Weeks Post-treatment: number analyzed (Participants) | 31 | 49
  4 Weeks Post-treatment | -1.8 [-5.00 to 1.30] | -0.6 [-2.00 to 0.80]

5. Other Pre Specified Outcome: Average Total Daily Duration of Medium Intensity Nosebleeds - Change From Baseline
Description: The daily of medium intensity epistaxis duration is calculated as the total duration of "dripping quickly" or "steady stream" nose bleeding events in a day, averaged across all days reported in a 4-week smartphone diary. The outcome is the change between the baseline diary on the specified timepoint
Time Frame: After 12 and 24 weeks of treatment, and 4 weeks post-treatment
Population: An intent-to-treat (ITT) analysis which included all randomized participants who provided outcome data.
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 43 | 73
minutes
  12 Weeks: number analyzed (Participants) | 35 | 64
  12 Weeks | -1.9 [-4.10 to 0.40] | -3.6 [-6.00 to -1.30]
  24 Weeks: number analyzed (Participants) | 32 | 53
  24 Weeks | -3.6 [-8.70 to 1.60] | -2.2 [-7.00 to 2.70]
  4 Weeks Post-treatment: number analyzed (Participants) | 31 | 49
  4 Weeks Post-treatment | -2 [-6.30 to 2.40] | -2.5 [-4.90 to 0.00]

6. Other Pre Specified Outcome: Average Total Daily Duration of High Intensity Nosebleeds - Change From Baseline
Description: The daily of high intensity epistaxis duration is calculated as the total duration of "gushing" or "pouring" nose bleeding events in a day, averaged across all days reported in a 4-week smartphone diary. The outcome is the change between the baseline diary on the specified timepoint
Time Frame: After 12 and 24 weeks of treatment, and 4 weeks post-treatment
Population: An intent-to-treat (ITT) analysis which included all randomized participants who provided outcome data.
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 43 | 73
minutes
  12 Weeks: number analyzed (Participants) | 35 | 64
  12 Weeks | -0.1 [-1.50 to 1.20] | -1.4 [-2.60 to -0.20]
  24 Weeks: number analyzed (Participants) | 32 | 53
  24 Weeks | 1.9 [-2.70 to 6.50] | -1.5 [-2.80 to -0.10]
  4 Weeks Post-treatment: number analyzed (Participants) | 31 | 49
  4 Weeks Post-treatment | 2 [-3.90 to 7.90] | -1.6 [-3.30 to 0.10]

7. Secondary Outcome: Total Iron Infused
Description: Total iron infused (mg) is calculated as the total in 4 weeks, averaged across all visits reported through the 24-week treatment period. Patients with no infusions have a value of zero.
Time Frame: Baseline through 24 Weeks
Population: An intent-to-treat (ITT) analysis which included all randomized participants who provided outcome data.
Measure: Median (Inter-Quartile Range); unit: mg/4 weeks
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 49 | 92
mg/4 weeks | 204 [33 to 341] | 170 [0 to 408]

8. Secondary Outcome: Total Iron Infused
Description: Total iron infused (mg) is calculated as the total in 4 weeks, averaged across all visits reported through the first 12 weeks of the treatment period. Patients with no infusions have a value of zero.
Time Frame: Baseline through 12 Weeks
Population: An intent-to-treat (ITT) analysis which included all randomized participants who provided outcome data.
Measure: Median (Inter-Quartile Range); unit: mg/4 weeks
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 49 | 92
mg/4 weeks | 170 [0 to 340] | 225 [0 to 510]

9. Secondary Outcome: Total Iron Infused
Description: Total iron infused (mg) is calculated as the total in 4 weeks, averaged across all visits reported through the second 12 weeks of the treatment period. Patients with no infusions have a value of zero.
Time Frame: 12 through 24 Weeks
Population: An intent-to-treat (ITT) analysis which included all randomized participants who provided outcome data.
Measure: Median (Inter-Quartile Range); unit: mg/4 weeks
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 45 | 74
mg/4 weeks | 333.3 [0 to 500] | 0 [0 to 340]

10. Secondary Outcome: Patients With Any Packed Red Blood Cells Transfusion Through 24 Weeks
Description: Patients with any packed red blood cells transfusion through the 24-week treatment period
Time Frame: Baseline through 24 Weeks
Population: An intent-to-treat (ITT) analysis which included all randomized participants who provided outcome data.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 49 | 92
Participants
  No transfusion | 38 | 77
  Yes transfusion | 11 | 15

11. Other Pre Specified Outcome: Total Blood Transfused
Description: Total blood transfused (units of blood) is calculated as the total in 4 weeks, averaged across all visits reported through the 24-week treatment period. Patients with no transfusions have a value of zero.
Time Frame: Baseline through 24 Weeks
Population: An intent-to-treat (ITT) analysis which included all randomized participants who provided outcome data.
Measure: Median (Inter-Quartile Range); unit: units of blood/4 weeks
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 49 | 92
units of blood/4 weeks | 0 [0.00 to 0.00] | 0 [0.00 to 0.00]

12. Secondary Outcome: Patients With Any Packed Red Blood Cells Transfusion Through 12 Weeks
Description: Patients with any packed red blood cells transfusion through the first 12 weeks of the treatment period
Time Frame: Baseline through 12 Weeks
Population: An intent-to-treat (ITT) analysis which included all randomized participants who provided outcome data.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 49 | 92
Participants
  No transfusion | 43 | 79
  Yes transfusion | 6 | 13

13. Other Pre Specified Outcome: Total Blood Transfused
Description: Total blood transfused (units of blood) is calculated as the total in 4 weeks, averaged across all visits reported through the first 12 weeks of the treatment period. Patients with no transfusions have a value of zero.
Time Frame: Baseline through 12 Weeks
Population: An intent-to-treat (ITT) analysis which included all randomized participants who provided outcome data.
Measure: Median (Inter-Quartile Range); unit: units of blood/4 weeks
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 49 | 92
units of blood/4 weeks | 0 [0.00 to 0.00] | 0 [0.00 to 0.00]

14. Secondary Outcome: Patients With Any Packed Red Blood Cells Transfusion 12-24 Weeks
Description: Patients with any packed red blood cells transfusion through the second 12 weeks of the treatment period
Time Frame: 12 through 24 Weeks
Population: An intent-to-treat (ITT) analysis which included all randomized participants who provided outcome data.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 45 | 74
Participants
  No transfusion | 37 | 67
  Yes transfusion | 8 | 7

15. Other Pre Specified Outcome: Total Blood Transfused
Description: Total blood transfused (units of blood) is calculated as the total in 4 weeks, averaged across all visits reported through the second 12 weeks of the treatment period. Patients with no transfusions have a value of zero.
Time Frame: 12 through 24 Weeks
Population: An intent-to-treat (ITT) analysis which included all randomized participants who provided outcome data.
Measure: Median (Inter-Quartile Range); unit: units of blood/4 weeks
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 45 | 74
units of blood/4 weeks | 0 [0.00 to 0.00] | 0 [0.00 to 0.00]

16. Other Pre Specified Outcome: Transferrin Saturation
Description: Change from baseline transferrin saturation collected from blood iron studies
Time Frame: After 4, 8, 12, 16, 20 and 24 weeks of treatment, and 4 weeks post-treatment
Population: An intent-to-treat (ITT) analysis which included all randomized participants who provided outcome data.
Measure: Mean (95% Confidence Interval); unit: Percent
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 49 | 87
Percent
  4 Weeks: number analyzed (Participants) | 46 | 84
  4 Weeks | 8.2 [-7.20 to 23.60] | -3.7 [-8.70 to 1.20]
  8 Weeks: number analyzed (Participants) | 45 | 77
  8 Weeks | 4.4 [-4.10 to 12.80] | -1.1 [-6.60 to 4.40]
  12 Weeks: number analyzed (Participants) | 42 | 70
  12 Weeks | -2.3 [-7.90 to 3.40] | 9 [-2.50 to 20.60]
  16 Weeks: number analyzed (Participants) | 39 | 62
  16 Weeks | 3.8 [-4.70 to 12.30] | 3.3 [-2.60 to 9.20]
  20 Weeks: number analyzed (Participants) | 42 | 59
  20 Weeks | 6.2 [-5.30 to 17.80] | 1.5 [-3.80 to 6.80]
  24 Weeks: number analyzed (Participants) | 39 | 58
  24 Weeks | 10.1 [-0.30 to 20.40] | 22.7 [-17.50 to 62.90]
  4 Weeks Post-treatment: number analyzed (Participants) | 36 | 56
  4 Weeks Post-treatment | 12.8 [-9.40 to 35.10] | 1.2 [-4.20 to 6.50]

17. Other Pre Specified Outcome: Ferritin
Description: Change from baseline ferritin level collected from blood iron studies
Time Frame: After 4, 8, 12, 16, 20 and 24 weeks of treatment, and 4 weeks post-treatment
Population: An intent-to-treat (ITT) analysis which included all randomized participants who provided outcome data.
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 49 | 92
ng/mL
  4 Weeks: number analyzed (Participants) | 49 | 88
  4 Weeks | -25.5 [-48.50 to -2.60] | -6.5 [-42.30 to 29.40]
  8 Weeks: number analyzed (Participants) | 48 | 83
  8 Weeks | 11.5 [-28.40 to 51.30] | 2.6 [-45.40 to 50.60]
  12 Weeks: number analyzed (Participants) | 45 | 75
  12 Weeks | -12.4 [-48.10 to 23.30] | 2.5 [-32.20 to 37.10]
  16 Weeks: number analyzed (Participants) | 42 | 69
  16 Weeks | 13.1 [-35.40 to 61.50] | 8.2 [-32.10 to 48.40]
  20 Weeks: number analyzed (Participants) | 42 | 62
  20 Weeks | 31.6 [-24.70 to 87.90] | -7.4 [-46.30 to 31.50]
  24 Weeks: number analyzed (Participants) | 42 | 61
  24 Weeks | 47.4 [-12.30 to 107.10] | -5.4 [-41.00 to 30.20]
  4 Weeks Post-treatment: number analyzed (Participants) | 38 | 62
  4 Weeks Post-treatment | -10.9 [-49.30 to 27.40] | -18.5 [-59.80 to 22.90]

18. Other Pre Specified Outcome: Hemoglobin
Description: Change from baseline Hemoglobin level taken from complete blood counts
Time Frame: After 4, 8, 12, 16, 20 and 24 weeks of treatment, and 4 weeks post-treatment
Population: An intent-to-treat (ITT) analysis which included all randomized participants who provided outcome data.
Measure: Mean (95% Confidence Interval); unit: g/dL
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 49 | 91
g/dL
  4 Weeks | -0.2 [-0.50 to 0.20] | -0.4 [-0.70 to -0.10]
  8 Weeks: number analyzed (Participants) | 48 | 85
  8 Weeks | -0.3 [-0.70 to 0.10] | -0.3 [-0.60 to 0.10]
  12 Weeks: number analyzed (Participants) | 45 | 75
  12 Weeks | 0 [-0.60 to 0.60] | 0 [-0.40 to 0.40]
  16 Weeks: number analyzed (Participants) | 43 | 71
  16 Weeks | -0.2 [-0.90 to 0.40] | 0.4 [-0.10 to 0.80]
  20 Weeks: number analyzed (Participants) | 44 | 65
  20 Weeks | 0 [-0.60 to 0.70] | 0.4 [-0.20 to 0.90]
  24 Weeks: number analyzed (Participants) | 42 | 62
  24 Weeks | -0.1 [-0.60 to 0.50] | 0.3 [-0.20 to 0.90]
  4 Weeks Post-treatment: number analyzed (Participants) | 40 | 62
  4 Weeks Post-treatment | -0.5 [-1.20 to 0.20] | 0.7 [0.10 to 1.20]

19. Other Pre Specified Outcome: Hematocrit
Description: Change from baseline Hematocrit level taken from complete blood counts
Time Frame: After 4, 8, 12, 16, 20 and 24 weeks of treatment, and 4 weeks post-treatment
Population: An intent-to-treat (ITT) analysis which included all randomized participants who provided outcome data.
Measure: Mean (95% Confidence Interval); unit: Percent
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 49 | 91
Percent
  4 Weeks | -0.3 [-1.40 to 0.80] | -1.4 [-2.30 to -0.40]
  8 Weeks: number analyzed (Participants) | 48 | 85
  8 Weeks | -0.7 [-1.90 to 0.50] | -0.9 [-2.10 to 0.30]
  12 Weeks: number analyzed (Participants) | 45 | 75
  12 Weeks | 0.1 [-1.40 to 1.60] | -0.2 [-1.50 to 1.10]
  16 Weeks: number analyzed (Participants) | 43 | 71
  16 Weeks | -0.6 [-2.40 to 1.20] | 0.4 [-1.00 to 1.70]
  20 Weeks: number analyzed (Participants) | 44 | 65
  20 Weeks | -0.3 [-2.00 to 1.40] | 0.2 [-1.30 to 1.70]
  24 Weeks: number analyzed (Participants) | 42 | 62
  24 Weeks | -0.7 [-2.30 to 0.90] | 0.3 [-1.30 to 1.90]
  4 Weeks Post-treatment: number analyzed (Participants) | 40 | 62
  4 Weeks Post-treatment | -1.6 [-3.50 to 0.30] | 1 [-0.40 to 2.40]

20. Other Pre Specified Outcome: Mean Corpuscular Volume (MCV)
Description: Change from baseline MCV level taken from complete blood counts
Time Frame: After 4, 8, 12, 16, 20 and 24 weeks of treatment, and 4 weeks post-treatment
Population: An intent-to-treat (ITT) analysis which included all randomized participants who provided outcome data.
Measure: Mean (95% Confidence Interval); unit: fL
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 49 | 91
fL
  4 Weeks | -0.1 [-1.10 to 0.80] | -0.4 [-1.30 to 0.40]
  8 Weeks: number analyzed (Participants) | 48 | 85
  8 Weeks | 0 [-1.10 to 1.10] | -1.2 [-2.30 to -0.20]
  12 Weeks: number analyzed (Participants) | 45 | 75
  12 Weeks | 0.1 [-1.30 to 1.40] | 0.1 [-1.00 to 1.20]
  16 Weeks: number analyzed (Participants) | 43 | 71
  16 Weeks | -0.2 [-2.00 to 1.60] | 0.9 [-0.40 to 2.10]
  20 Weeks: number analyzed (Participants) | 44 | 65
  20 Weeks | 1.3 [-0.60 to 3.20] | 2.2 [0.70 to 3.60]
  24 Weeks: number analyzed (Participants) | 42 | 62
  24 Weeks | 1.6 [-0.50 to 3.70] | 3.2 [1.60 to 4.80]
  4 Weeks Post-treatment: number analyzed (Participants) | 38 | 62
  4 Weeks Post-treatment | 0.2 [-1.80 to 2.30] | 3.2 [1.60 to 4.70]

21. Other Pre Specified Outcome: Mean Corpuscular Hemoglobin Concentration (MCHC)
Description: Change from baseline MCHC level taken from complete blood counts
Time Frame: After 4, 8, 12, 16, 20 and 24 weeks of treatment, and 4 weeks post-treatment
Population: An intent-to-treat (ITT) analysis which included all randomized participants who provided outcome data.
Measure: Mean (95% Confidence Interval); unit: g/dL
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 47 | 91
g/dL
  4 Weeks: number analyzed (Participants) | 47 | 89
  4 Weeks | -0.2 [-0.50 to 0.10] | 0 [-0.30 to 0.30]
  8 Weeks: number analyzed (Participants) | 46 | 85
  8 Weeks | -0.2 [-0.50 to 0.10] | 0.1 [-0.20 to 0.40]
  12 Weeks: number analyzed (Participants) | 43 | 75
  12 Weeks | 0 [-0.50 to 0.40] | 0.1 [-0.20 to 0.40]
  16 Weeks: number analyzed (Participants) | 42 | 71
  16 Weeks | -0.2 [-0.70 to 0.30] | 0.6 [0.30 to 1.00]
  20 Weeks: number analyzed (Participants) | 43 | 65
  20 Weeks | 0.3 [-0.30 to 0.90] | 0.7 [0.30 to 1.20]
  24 Weeks: number analyzed (Participants) | 41 | 62
  24 Weeks | 0 [-0.40 to 0.40] | 0.6 [0.20 to 1.10]
  4 Weeks Post-treatment: number analyzed (Participants) | 38 | 62
  4 Weeks Post-treatment | -0.2 [-0.70 to 0.30] | 0.9 [0.30 to 1.40]

22. Other Pre Specified Outcome: Platelets
Description: Change from baseline platelets taken from complete blood counts
Time Frame: After 4, 8, 12, 16, 20 and 24 weeks of treatment, and 4 weeks post-treatment
Population: An intent-to-treat (ITT) analysis which included all randomized participants who provided outcome data.
Measure: Mean (95% Confidence Interval); unit: 10^3/uL platelets
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 49 | 91
10^3/uL platelets
  4 Weeks | 7.8 [-5.70 to 21.30] | 13.4 [-8.00 to 34.90]
  8 Weeks: number analyzed (Participants) | 47 | 85
  8 Weeks | -2.3 [-17.40 to 12.70] | 19.3 [-0.60 to 39.20]
  12 Weeks: number analyzed (Participants) | 44 | 75
  12 Weeks | 4.9 [-12.90 to 22.70] | 0.9 [-18.20 to 20.10]
  16 Weeks: number analyzed (Participants) | 43 | 71
  16 Weeks | 10.3 [-15.90 to 36.50] | -19.7 [-36.90 to -2.50]
  20 Weeks: number analyzed (Participants) | 44 | 65
  20 Weeks | -2.1 [-18.10 to 13.90] | -24.1 [-46.10 to -2.10]
  24 Weeks: number analyzed (Participants) | 42 | 62
  24 Weeks | 4 [-11.50 to 19.50] | -27.3 [-51.50 to -3.00]
  4 Weeks Post-treatment: number analyzed (Participants) | 38 | 61
  4 Weeks Post-treatment | 5.7 [-11.60 to 22.90] | -13 [-33.00 to 7.00]

23. Secondary Outcome: Neuro-QoL - Satisfaction With Social Roles and Activities - T Score
Description: The outcome measure is the Neuro-QoL Satisfaction with Social Roles and Activities T-Score to compare the outcomes of Pomalidomide versus Placebo. The Neuro-QoL Satisfaction with Social Roles and Activities Short Form (V1.1) T-score has a value of 50 representing the average general US population, with a standard deviation of 10, and with higher scores indicating more satisfaction. The minimal detectable change is 3.7 T score points
Time Frame: Baseline, after 12 and 24 weeks of treatment, and 4 weeks post-treatment
Population: An intent-to-treat (ITT) analysis which included all randomized participants who provided outcome data.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 48 | 92
units on a scale
  Baseline: number analyzed (Participants) | 48 | 91
  Baseline | 44.7 [42.9 to 46.4] | 45.5 [44.1 to 46.8]
  12 Weeks: number analyzed (Participants) | 43 | 71
  12 Weeks | 46.5 [44.6 to 48.4] | 47.5 [46.1 to 49.0]
  24 Weeks: number analyzed (Participants) | 41 | 59
  24 Weeks | 46 [43.7 to 48.2] | 47.6 [46.0 to 49.3]
  4 Weeks Post-treatment: number analyzed (Participants) | 37 | 71
  4 Weeks Post-treatment | 45.6 [43.0 to 48.3] | 48.8 [47.2 to 50.4]

24. Secondary Outcome: Patient Reported Outcomes Measurement Information System (PROMIS) - Emotional Distress - Depression - T Score
Description: The outcome measure is the PROMIS Emotional Distress - Depression T-Score to compare the outcomes of Pomalidomide versus Placebo. The PROMIS Emotional Distress-Depression Short Form (V1.0) T-score has a value of 50 representing the average general US population, with a standard deviation of 10, and with higher scores indicating more depression
Time Frame: Baseline, after 12 and 24 weeks of treatment, and 4 weeks post-treatment
Population: An intent-to-treat (ITT) analysis which included all randomized participants who provided outcome data.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 49 | 92
units on a scale
  Baseline: number analyzed (Participants) | 49 | 91
  Baseline | 0.2 [0.00 to 0.50] | -0.1 [-0.30 to 0.10]
  12 Weeks: number analyzed (Participants) | 44 | 71
  12 Weeks | 0 [-0.30 to 0.30] | -0.1 [-0.30 to 0.10]
  24 Weeks: number analyzed (Participants) | 42 | 59
  24 Weeks | -0.1 [-0.40 to 0.20] | -0.2 [-0.40 to 0.10]
  4 Weeks Post-treatment: number analyzed (Participants) | 37 | 72
  4 Weeks Post-treatment | 0.1 [-0.30 to 0.50] | -0.3 [-0.50 to -0.10]

25. Secondary Outcome: PROMIS - Fatigue - T Score
Description: The outcome measure is the PROMIS Fatigue T-Score to compare the outcomes of Pomalidomide versus Placebo. The PROMIS® Fatigue Short Form (V1.0) T-score has a value of 50 representing the average general US population, with a standard deviation of 10, and with higher scores indicating more fatigue
Time Frame: Baseline, after 12 and 24 weeks of treatment, and 4 weeks post-treatment
Population: An intent-to-treat (ITT) analysis which included all randomized participants who provided outcome data.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 49 | 92
units on a scale
  Baseline: number analyzed (Participants) | 49 | 91
  Baseline | 57.7 [54.6 to 60.8] | 55.7 [53.6 to 57.8]
  12 Weeks: number analyzed (Participants) | 44 | 71
  12 Weeks | 55.8 [53.2 to 58.3] | 54.7 [52.5 to 56.9]
  24 Weeks: number analyzed (Participants) | 42 | 59
  24 Weeks | 56.2 [52.9 to 59.6] | 54.2 [51.6 to 56.9]
  4 Weeks Post-treatment: number analyzed (Participants) | 37 | 72
  4 Weeks Post-treatment | 59.5 [56.0 to 63.1] | 52.3 [50.1 to 54.5]

26. Secondary Outcome: HHT-Specific QOL Questionnaire - Score
Description: The outcome measure is the HHT-Specific QOL Questionnaire - Score to compare the outcomes of Pomalidomide versus Placebo. The HHT-specific QOL score ranges from 0 to 16 with higher scores indicating more limitations due to HHT in the prior 4 weeks
Time Frame: Baseline, after 12 and 24 weeks of treatment, and 4 weeks post-treatment
Population: An intent-to-treat (ITT) analysis which included all randomized participants who provided outcome data.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Pomalidomide
Number analyzed (Participants) | 49 | 91
units on a scale
  Baseline: number analyzed (Participants) | 48 | 90
  Baseline | 7.1 [6.10 to 8.10] | 5.8 [5.20 to 6.40]
  12 Weeks: number analyzed (Participants) | 44 | 70
  12 Weeks | 5 [3.90 to 6.10] | 3.5 [2.70 to 4.30]
  24 Weeks: number analyzed (Participants) | 42 | 59
  24 Weeks | 5.6 [4.40 to 6.80] | 3.6 [2.80 to 4.30]
  4 Weeks Post-treatment: number analyzed (Participants) | 37 | 72
  4 Weeks Post-treatment | 5.9 [4.50 to 7.40] | 3.7 [2.90 to 4.40]

ADVERSE EVENTS:
Time Frame: 6 Months
Description: Patients were randomized to 2 groups: placebo and pomalidomide. All patients in the pomalidomide group were started on 4 mg and dose could be reduced (to 3 mg or 2 mg) or temporarily stopped by the investigator due to side effects. So a single participant could have administrations of each of the 4 mg, 3 mg, and 2 mg doses during the course of the study.
  Since participants were not necessarily unique to a dose level, adverse events are presented by treatment and not by treatment and dose.
Arm/Group | Placebo | Pomalidomide
All-Cause Mortality (participants affected / at risk) | 0/49 | 1/95
Serious Adverse Events (participants affected / at risk) | 8/49 | 22/95
Other Adverse Events (participants affected / at risk) | 43/49 | 90/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=49) | Pomalidomide (N=95)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (2)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Arteriovenous malformation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (4) | 1 (2)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Corona virus infection (Infections and infestations) | 0 (0) | 1 (1)
Extradural abscess (Infections and infestations) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1)
Liver abscess (Infections and infestations) | 0 (0) | 1 (1)
Pilonidal cyst (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 2 (2)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Cardiac ablation (Surgical and medical procedures) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=49) | Pomalidomide (N=95)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Increased tendency to bruise (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 5 (5)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 9 (15)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 5 (9) | 41 (70)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 4 (6)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure high output (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac hypertrophy (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac valve disease (Cardiac disorders) | 0 (0) | 1 (1)
Cardiomegaly (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 2 (2)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 3 (3)
Tricuspid valve incompetence (Cardiac disorders) | 1 (1) | 1 (1)
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Hepatic arteriovenous malformation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Ichthyosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Otorrhoea (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 2 (2)
Blepharitis (Eye disorders) | 0 (0) | 1 (1)
Corneal scar (Eye disorders) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 2 (2)
Eye irritation (Eye disorders) | 1 (1) | 2 (2)
Eye pruritus (Eye disorders) | 0 (0) | 1 (1)
Ulcerative keratitis (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 8 (8)
Abdominal pain (Gastrointestinal disorders) | 3 (4) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 3 (3)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 9 (9) | 45 (51)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 7 (8)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 9 (9)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Faeces discoloured (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric polyps (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal angiectasia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 1 (1) | 1 (2)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Glossodynia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lip dry (Gastrointestinal disorders) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 8 (8) | 15 (16)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral dysaesthesia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retching (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Splenic artery aneurysm (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tongue eruption (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tongue haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 4 (4)
Asthenia (General disorders) | 0 (0) | 2 (2)
Chest discomfort (General disorders) | 0 (0) | 2 (2)
Chest pain (General disorders) | 0 (0) | 2 (2)
Chills (General disorders) | 0 (0) | 3 (3)
Discomfort (General disorders) | 0 (0) | 1 (1)
Face oedema (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 17 (20) | 42 (48)
Feeling abnormal (General disorders) | 1 (1) | 1 (1)
Feeling jittery (General disorders) | 0 (0) | 1 (1)
Generalised oedema (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 3 (3)
Localised oedema (General disorders) | 1 (1) | 0 (0)
Loss of control of legs (General disorders) | 0 (0) | 1 (1)
Mucosal dryness (General disorders) | 0 (0) | 2 (2)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Oedema (General disorders) | 1 (1) | 5 (5)
Oedema peripheral (General disorders) | 1 (1) | 14 (14)
Pain (General disorders) | 1 (1) | 4 (4)
Pyrexia (General disorders) | 1 (1) | 3 (3)
Sensation of foreign body (General disorders) | 0 (0) | 1 (1)
Thirst (General disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hepatic lesion (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 3 (3)
Multiple allergies (Immune system disorders) | 0 (0) | 2 (2)
Seasonal allergy (Immune system disorders) | 1 (1) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2)
Bursitis infective (Infections and infestations) | 0 (0) | 1 (1)
Carbuncle (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1)
Corona virus infection (Infections and infestations) | 9 (9) | 9 (9)
Eye infection (Infections and infestations) | 0 (0) | 1 (1)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1)
Infective glossitis (Infections and infestations) | 1 (2) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Lip infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 4 (4)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (3) | 3 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 5 (6)
Viral pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Radiation skin injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vaccination complication (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (2)
Cardiac murmur (Investigations) | 2 (2) | 2 (2)
Heart rate increased (Investigations) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1)
Right ventricular systolic pressure increased (Investigations) | 0 (0) | 1 (1)
Weight increased (Investigations) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (3) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 (7) | 13 (14)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Focal nodular hyperplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Anosmia (Nervous system disorders) | 0 (0) | 1 (1)
Disturbance in attention (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 7 (8) | 16 (17)
Dysgeusia (Nervous system disorders) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 3 (5) | 13 (14)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 3 (3) | 0 (0)
Hypogeusia (Nervous system disorders) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 3 (3)
Mental impairment (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 2 (2)
Paraesthesia (Nervous system disorders) | 2 (3) | 4 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 2 (2)
Somnolence (Nervous system disorders) | 2 (2) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 2 (2)
Tremor (Nervous system disorders) | 0 (0) | 8 (8)
Anxiety (Psychiatric disorders) | 1 (1) | 3 (3)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 5 (5) | 4 (4)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 3 (3)
Renal cyst (Renal and urinary disorders) | 2 (2) | 0 (0)
Breast tenderness (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Menstruation irregular (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Scrotal oedema (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Scrotal swelling (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 22 (24)
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 6 (6)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Palmar erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 13 (14)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 20 (20)
Rash erythematous (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (6)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin warm (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 6 (7)
Cataract operation (Surgical and medical procedures) | 0 (0) | 1 (2)
Gastrointestinal endoscopic therapy (Surgical and medical procedures) | 1 (1) | 0 (0)
Sinus operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 1 (1) | 0 (0)
Transurethral bladder resection (Surgical and medical procedures) | 0 (0) | 1 (1)
Angiopathy (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Fibromuscular dysplasia (Vascular disorders) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 3 (3)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Pallor (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1)
Varicose vein ruptured (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (4):
  • Study Protocol (2022-09-30): https://cdn.clinicaltrials.gov/large-docs/44/NCT03910244/Prot_004.pdf
  • Statistical Analysis Plan (2023-09-28): https://cdn.clinicaltrials.gov/large-docs/44/NCT03910244/SAP_001.pdf
  • Informed Consent Form: Part 1 Master Consent (2022-10-25): https://cdn.clinicaltrials.gov/large-docs/44/NCT03910244/ICF_002.pdf
  • Informed Consent Form: Part 2 Local Site Information Consent (2020-03-09): https://cdn.clinicaltrials.gov/large-docs/44/NCT03910244/ICF_003.pdf